CLINICAL TRIAL: NCT05815485
Title: A Randomized, Double-Blind, Placebo-Controlled Phase 2/3 Study to Determine the Safety and Effectiveness of Azeliragon in the Treatment of Patients Hospitalized for Coronavirus Disease 2019 (COVID-19) or Pneumonia
Status: Active, not recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: The University of Texas Medical Branch, Galveston (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 24-0103; HUM00221960 (Other: University of Michigan)
Record Dates: First submitted 2023-04-13; First posted 2023-04-18 (Actual); Last update posted 2025-03-03 (Actual); Status verified 2025-02

CONDITIONS: COVID-19
Keywords: Azeliragon; Acute Kidney Injury
MeSH Terms: conditions — COVID-19; Acute Kidney Injury | interventions — azeliragon

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Azeliragon and placebo will be dispensed and labeled by the unblinded research pharmacist at each site in a blinded manner that will not reveal if the product dispensed is active or placebo.
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Phase 2 azeliragon (Experimental)
  Interventions: Drug: Azeliragon
- Phase 2 placebo (Placebo Comparator)
  Interventions: Drug: Placebo
- Phase 3 azeliragon (Experimental)
  Interventions: Drug: Azeliragon
- Phase 3 placebo (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azeliragon — 30 mg twice daily for 5 days followed by 20 mg once daily for 5 days or until discharge (whichever is earliest).
  Arms: Phase 2 azeliragon; Phase 3 azeliragon
Drug: Placebo — Twice daily for 5 days then 1 time daily for 5 days or until discharge (whichever is earliest).
  Arms: Phase 2 placebo; Phase 3 placebo

SUMMARY:
A new drug called azeliragon could be used to treat patients with COVID-19 or other pneumonia infections but the researchers don't know. In this study, they are learning the effects of azeliragon patients hospitalized for COVID-19 or pneumonia.

ELIGIBILITY:
Inclusion Criteria:

* Patients with at least two of the following signs or symptoms: cough, chest pain, shortness of breath, hypoxia (oxygen saturation <90%)
* Clinical diagnosis of pneumonia or COVID-19 during the first 48 hours of hospitalization.
* Patients admitted to the hospital within the previous 48 hours (from time of admission to initial treatment dose.)
* Provide informed consent to participate in the study (by participant or legally-acceptable representative).

Exclusion Criteria:

* Patients for whom intubation within 24 hours of admission is considered likely.
* Alanine aminotransferase (ALT) or aspartate aminotransferase (AST) >3x upper limit of normal (ULN), OR total serum bilirubin >2x ULN.
* Patients who were receiving dialysis as a regular treatment at the time of admission. (Participants are not excluded for historic need for dialysis.)
* Chronic liver disease with Child-Pugh class B of (7 to 9) or higher.
* Patients with an electrocardiogram (ECG) corrected QT interval (QTc) > 500 ms.
* Patients requiring treatment with strong inhibitors of CYP2C8
* Females of childbearing potential who are pregnant, breastfeeding, and/or not using a highly-effective method of contraception (consistent with local regulations regarding the methods of contraception for those participating in clinical studies, including willingness to use 2 acceptable forms of contraception from screening until after the end of drug treatment. Acceptable forms include tubal ligation, male latex condom with or without spermicide, partner's vasectomy, diaphragm with spermicide, intrauterine device, cervical cap/sponge with spermicide, contraceptive sponge, female condom, hormonal contraceptive including oral, transdermal, vaginal ring, subcutaneous injection, or implanted rod.)
* Allergy to azeliragon or formulation excipients in the azeliragon or placebo capsule.
* Concurrent participation in another device or drug trial for treatment purposes. Trials with devices intended for diagnostic purposes only are allowable..
* Any other condition, including abnormal laboratory values that, in the judgment of the investigator, could put the participant at increased risk, or would interfere with the conduct or planned analysis of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2023-05-04 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-04 (Estimated)

PRIMARY OUTCOMES:
Frequency of Adverse Events (AEs) (Phase 2 only) | Up to 28 days post-treatment
  Including overall, treatment-related, Grade 3 or higher in severity, serious AEs (SAEs), fatal, and those resulting in treatment discontinuation
Death, need for mechanical ventilation or Acute Kidney Injury (AKI) of stage 2 or higher per Kidney Disease Improving Global Outcomes (KDIGO) scale (Phase 3 only) | Day 14 of hospitalization
  The primary outcome is a composite endpoint, which is defined as the need for mechanical ventilation, in-hospital death or AKI of stage 2 or higher per KDIGO scale.
  There are 3 stages in the KDIGO scale with stage 3 being the worst (corresponds to renal failure).
  KDIGO Scale definitions: Stage 2 - Serum Creatinine 2-2.9 times baseline Stage 3 - Serum Creatinine 3 times baseline or Increase in serum creatinine to ≥4 mg/dL or Initiation of renal replacement therapy

SECONDARY OUTCOMES:
Frequency of each AKI Kidney Disease Improving Global Outcomes (KDIGO) scale scores (Phase 3 only) | Day 14 of hospitalization
  There are 3 stages in the KDIGO scale with stage 3 being the worst (corresponds to renal failure).
  Stage 1- serum creatinine 1.5 to 1.9 times baseline OR an increase in serum creatinine ≥ 0.3 mg/dL OR urine output < 0.5ml/kg/hour for 6-12 hours. Stage 2- serum creatinine 2.0-2.9 times baseline OR urine output <0.5mg/kg/hour for ≥ 12 hours Stage 3- serum creatinine 3.0 times baseline (or serum creatinine of more than or equal to 4.0 mg/dl with an acute increase of at least 0.5 mg/dl) (OR) Urine output less than 0.3 ml/kg/hour for 24 hours or anuria for 12 hours or new renal replacement therapy
Frequency of sustained renal function (Phase 3 only) | Day 14 of hospitalization
  Renal function defined by no increase in serum creatinine of ≥0.3mg/dL during any 48hr period, AND no increase in serum creatinine of ≥1.5 times
Frequency of renal function after prior AKI of stage 2 or higher (Phase 3 only) | Day 14 of hospitalization
  Serum creatinine levels to < 1.5 times baseline level
Frequency of Intensive Care Unit (ICU) admission (Phase 3 only) | Day 14 of hospitalization
Number of days in ICU (Phase 3 only) | Day 14 of hospitalization
Frequency of AEs (Phase 3 only) | Day 14 of hospitalization
  Including: overall, treatment-related, Grade 3 or higher in severity, serious, fatal, and those resulting in treatment discontinuation
Length of hospitalization (Phase 3 only) | Up to 14 days

CONTACTS AND LOCATIONS:
Overall Officials: Lucas S. Blanton, MD, Principal Investigator — University of Texas
Locations (3):
- United States (3):
  - Rush University, Chicago, Illinois
  - University of Michigan, Ann Arbor, Michigan
  - University of Texas Medical Branch, Galveston, Texas

IPD SHARING:
Plan to Share IPD: No